CLINICAL TRIAL: NCT07350928
Title: A Phase III Randomized Controlled Clinical Trial Evaluating the Efficacy of Preoperative Dexmedetomidine Hydrochloride Nasal Spray in Optimizing Awake Sedation During Breast-Conserving Surgery for Breast Cancer and Postoperative Awake Status
Brief Title: Observation of the Effect of Preoperative Use of Dexmedetomidine Hydrochloride Nasal Spray on Optimizing Awake Sedation During Breast-Conserving Surgery for Breast Cancer and Postoperative Awake Status
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yajing Yuan, Associate Chief Physician, Tianjin Medical University Cancer Institute and Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E20250012
Record Dates: First submitted 2025-12-15; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Induction of anesthesia with placebo spray prior to surgery (Placebo Comparator)
  Interventions: Drug: Induction of anesthesia with placebo spray prior to surgery
- Induction of anesthesia with dexmedetomidine nasal spray prior to surgery (Experimental)
  Interventions: Drug: Induction of anesthesia with dexmedetomidine nasal spray prior to surgery

INTERVENTIONS:
Drug: Induction of anesthesia with dexmedetomidine nasal spray prior to surgery — Induction of anesthesia with dexmedetomidine nasal spray prior to surgery
  Arms: Induction of anesthesia with dexmedetomidine nasal spray prior to surgery
Drug: Induction of anesthesia with placebo spray prior to surgery — Induction of anesthesia with placebo spray prior to surgery
  Arms: Induction of anesthesia with placebo spray prior to surgery

SUMMARY:
This clinical trial aims to evaluate the efficacy and safety of Dexmedetomidine Hydrochloride Nasal Spray for conscious sedation and anxiety relief during breast-conserving surgery. The main questions it aims to answer are:

Does Dexmedetomidine Hydrochloride Nasal Spray effectively provide intraoperative sedation and improve postoperative awakening time? What changes in vital signs or postoperative complications do participants experience when using this medication?

Researchers will compare Dexmedetomidine Hydrochloride Nasal Spray to a placebo (saline nasal spray) to determine its efficacy in breast-conserving surgery.

Participants will:

Receive preoperative administration of either Dexmedetomidine Hydrochloride Nasal Spray or the placebo nasal spray; Undergo regular intraoperative and postoperative assessments, including sedation scores, awakening time, and pain scores; Provide satisfaction feedback and be monitored for changes in vital signs and complications.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent for
* The patients included in the study were women aged between 20 and 70.
* ASA (American Society of Anesthesiologists) I-II.
* BMI:18-26 Kg/m ²

Exclusion Criteria:

* Subjects deemed unsuitable for nasal spray administration by the researchers (such as those with severe rhinitis, nasal deformities, etc.);
* Severe bradycardia (HR < 50 beats/min), history of cardiac conduction block;
* History of upper respiratory tract infection;
* History of asthma;
* History of allergy to DEX or local anesthetics;
* Subjects who have taken anti-anxiety medication before the operation;
* Subjects with a history of ischemic stroke or transient ischemic attack;
* Subjects with poorly controlled blood pressure despite medication;
* Subjects with a history of mental illness, cognitive impairment, or epilepsy;
* Subjects with a history of pregnancy;
* Subjects who have been taking sedatives or analgesics for a long time;
* Subjects with a history of liver or kidney function impairment;
* Subjects with a history of drug or alcohol abuse;
* Other situations that the reviewers consider to be disqualifying based on the registration study, such as potential non-compliance with the clinical protocol.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Observer's Assessment of Alterness/Sedation and Numerical rating scale | From enrollment to the end of the first postoperative day
  Used to assess the depth of patient sedation or anesthesia. This scale is primarily applied during surgery, intensive care, or sedation therapy. By observing indicators such as behavioral responses, facial expressions, and limb movements, it categorizes sedation levels into five grades (1-5 points). This aids healthcare providers in real-time monitoring and adjustment of sedation protocols to ensure safety and efficacy. By evaluating sedation scores, the sedative effect of dexmedetomidine hydrochloride can be quantified to determine whether it provides adequate sedation during surgery, ensuring patient comfort and cooperation.
Hospital Anxiety and Depression Scale (HADS) | From enrollment to the end of the first postoperative day
  The HADS is a commonly used tool for assessing patients' anxiety and depression, particularly in hospital settings. This scale consists of seven anxiety items and seven depression items, designed for rapid screening of anxiety and depression symptoms in patients.
  Scale Structure:
  Anxiety Section (HADS-A): 7 items, assessing patients' anxiety. Depression Section (HADS-D): 7 items, assessing patients' depression.
  Scoring Method:
  Each item is scored 0-3 points, yielding a total score range of 0-21 points. Higher scores indicate greater severity of anxiety or depression.
  0-7 points: Normal 8-10 points: Mild 11-14 points: Moderate 15 points and above: Severe HADS can screen patients' anxiety and depression status prior to medication administration, assisting healthcare providers in developing appropriate psychological intervention measures.

SECONDARY OUTCOMES:
Heart rate | From enrollment to the end of the first postoperative day
Patient and Surgeon Satisfaction Scores | From enrollment to the end of the first postoperative day
  Measurement Method: Patients and surgeons are each asked to rate the effectiveness of anesthesia and intraoperative sedation.
Pain Rating (VAS Visual Analog Scale) | From enrollment to the end of the first postoperative day
  Use the Visual Analogue Scale (VAS) to assess pain intensity at different postoperative time points.
  Visual Analogue Scale (VAS) 0 points: No pain 1-3 points: Mild pain 4-6 points: Moderate pain 7-10 points: Severe pain
Incidence of adverse reactions | From enrollment to the end of the first postoperative day
Restore quality assessment | From enrollment to the end of the first postoperative day
  Using the Quality of Recovery (QOR) Questionnaire Content: Assesses aspects including fatigue, pain, emotional state, and functional recovery. The scale ranges from 0 to 100 points, with higher scores indicating better recovery quality.
blood pressure | From enrollment to the end of the first postoperative day
respiratory rate | From enrollment to the end of the first postoperative day
oxygen saturation | From enrollment to the end of the first postoperative day

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No